CLINICAL TRIAL: NCT00604474
Title: Development of Auditory Skills in Young Deaf Children With Bilateral Cochlear Implants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not sufficient enrollment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07030750; ACR0906
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Deafness
Keywords: Deafness; Hearing Loss; Cochlear Implants; Advanced Bionics; HiResolution Bionic Ear System
MeSH Terms: conditions — Deafness; Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Device: HiResolution Bionic Ear System (Cochlear Implant)

INTERVENTIONS:
Device: HiResolution Bionic Ear System (Cochlear Implant) — Subjects are required to have bilateral implantation of the Advanced Bionics HiResolution Bionic Ear System (Cochlear Implant)

SUMMARY:
The primary objective to this study is to describe the auditory development and performance of young deaf children who receive bilateral implants during the first two years following device activation.

DETAILED DESCRIPTION:
The primary purpose of this study is to track patient outcomes for bilateral cochlear implant recipients in a cohort of children, ages 12 to 36 months at time of surgery, who receive two implants in the same operation or in two different surgeries with the initial fitting of the devices separated by no more than six months. Acquisition of auditory milestones and speech recognition skills, which underpin the development of spoken language, will be assessed on a battery of outcome measures typically used to quantify implant benefits. In addition, global quality of life and communicative performance will be assessed by parental proxy. Performance will be tracked after 3, 6, 12, 18, and 24 months of device use. The study also will identify variables that may predict the degree of bilateral implant benefit in young children (e.g., age at implant, pre-implant hearing thresholds, communication mode, family socioeconomic status, post-implant aided thresholds, simultaneous vs. staged placement of devices).

ELIGIBILITY:
Inclusion Criteria:

* Profound bilateral hearing loss (PTA>= 90dB HL)
* Have independently elected to undergo bilateral implantation of Advanced Bionics HiResolution Bionic Ear System and meet all the eligibility criteria for this device as described in the product labeling.
* Age at implant: 12-36 months
* Negligible benefit from hearing aids, defined as failure to reach developmentally appropriate milestones on IT-MAIS
* No previous cochlear implant use
* Normal/patent cochlea with no more than a mild "partitioning" defect in either ear
* English as the primary language spoken in the home
* Parental willingness to follow study protocol

Exclusion Criteria:

* Deafness secondary to meningitis
* Presence of other conditions that could affect performance on outcome measures or otherwise confound or interfere with study participation of outcomes measures.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Subject performance on speech perception tests | Two years post device activation

SECONDARY OUTCOMES:
Speech recognition performance at various intervals. Global quality of life and functional communicative performance completed by parental proxy | 3, 6, 12, 18, and 24 months post device activation

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lustig, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States